CLINICAL TRIAL: NCT03063957
Title: Identification and Characterization of Microbial and Immunologic Changes in Microscopic Colitis
Brief Title: Identification/Characterization of Changes in Microscopic Colitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry); American College of Gastroenterology (Other)
Responsible Party: Principal Investigator, Hamed Khalili, Assistant Professor of Medicine at Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2015P001333
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Colitis, Microscopic
MeSH Terms: conditions — Colitis, Microscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Microscopic Colitis: Patients with confirmed microscopic colitis
- Control: Patients that are not diagnosed with microscopic colitis

SUMMARY:
The goal of this study is to establish a prospective observational cohort of adult patients with microscopic colitis and collect clinical information and specimens over the course of their treatment. This information will be used in order to establish a patient registry with detailed clinical data and a specimen repository for future research as well as to specifically identify genetic and molecular characteristics associated with microscopic colitis.

DETAILED DESCRIPTION:
Microscopic colitis (MC) is a chronic relapsing disease of the colon, characterized by watery non-bloody diarrhea, usually normal colonoscopic findings, and typical histology findings. It is frequently accompanied by abdominal pain, nocturnal diarrhea, and mild weight loss. The incidence of MC has increased significantly over recent years with a 2010 study reporting U.S. incidence for MC as 19.7 per 100,000 person-years. MC comprises two major histological subtypes: collagenous colitis (CC), characterized by a distinctive thickened band of subepithelial collagen (>10-20um), and lymphocytic colitis (LC), with an increased number of intraepithelial lymphocytes (>20 lymphocytes per 100 epithelial cells).

Although the exact etiology of MC remains largely unknown, a few observational studies have suggested associations with autoimmune disorders (e.g. celiac disease, and thyroid disorders), cigarette smoking status, and medications such as non-steroidal anti-inflammatory drugs (NSAIDS), proton pump inhibitors (PPIs), selective serotonin reuptake inhibitors (SSRI), and statins. In addition to environmental factors, recently studies indicate that genetics and specific infectious organisms may also play a role in development of the disease. A recent study revealed a seasonal incidence pattern of lymphocytic colitis, suggesting a potential link to an infectious or allergic component. Further, one study demonstrated an association between collagenous colitis and persistent colonic C. difficile infection. Additionally, while familial occurrence of MC has been reported, suggesting a genetic predisposition, the roles of specific genetic factors have not been described. Finally, recent studies demonstrate an association between MC and various autoimmune disorders including celiac disease, autoimmune thyroid disease, and Sjören's syndrome, indicating that MC may be part of a broader spectrum of autoimmune disorders. Despite these findings, few studies have investigated the role of genetic, infectious, and immunological factors in the development and progression of MC.

Budesonide is the only treatment for MC that appeared to be effective in randomized controlled trials, with remission rates of 80%. However, recurrence of clinical symptoms following withdrawal of treatment is not uncommon. Thus, further investigation of the molecular mechanisms underlying MC is needed in order to obtain targeted and sustainable treatment.

Analysis of clinical specimens obtained by colonoscopy from individuals affected with MC over the course of their treatment offers a promising method by which to improve our understanding of MC. Profiling of genetic and molecular characteristics such as changes in gut flora, colonic mucosal immune profiles, and genetic factors over the course of treatment would provide powerful insight into the role of these factors in the pathophysiology of the disease which may ultimately lead to better treatments. Additionally, identification of disease biomarkers can aid in developing disease monitoring and surveillance strategies.

Here, we propose to establish a cohort of individuals with suspected microscopic colitis undergoing diagnostic colonoscopy at the Massachusetts General Hospital (MGH) to identify genetic and molecular characteristics associated with the progression of this disease. This study will elaborate on findings from a medical record review of patients with microscopic colitis treated at MGH from 2002 to 2014. In addition to medical records, genetic and molecular characteristics of colonic samples will be examined to determine their influence on treatment response and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Ability and willingness to comply with all patient visits and study-related procedures
* Ability to understand and complete all study-related materials and questionnaires
* Patients ages 18 or older with suspected microscopic colitis
* Patients that have been previously treated for microscopic colitis that are being seen for possible relapse will also be included

Exclusion Criteria:

* Inability to provide informed consent
* Inability or unwillingness to comply with all patient visits and study-related procedures
* Inability to understand and complete all study-related materials and questionnaires
* Patients with a known diagnosis of Inflammatory Bowel Disease or colorectal cancer
* Patients with a known bleeding disorder, acute disease, or those that are awaiting transplantation
* Patients who have taken antibiotics in the last two weeks
* Female subjects who are pregnant or nursing

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or established microscopic colitis who are scheduled to receive a diagnostic colonoscopy or attend an office visit at the MGH Gastroenterology Unit will be eligible for recruitment
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2015-06-30 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome Analysis | 1.5 years
  Standard 16s rRNA sequencing for taxonomic identification and metagenomic profiling of the gut microbiome will be performed on stool and tissue samples.
Immune Response | 1.5 years
  Immune cells in blood and biopsy samples will be sorted and quantified using flow cytometry

SECONDARY OUTCOMES:
α4β7 in microscopic colitis pathogenesis | 2 years
  Vedolizumab will be used as a reagent for in vitro identification and investigation of eosinophils that express α4β7

CONTACTS AND LOCATIONS:
Overall Officials: Hamed Khalili, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified information may be shared with other collaborators and entities involved in generating data.

REFERENCES:
- [Background] Brown WR, Tayal S. Microscopic colitis. A review. J Dig Dis. 2013 Jun;14(6):277-81. doi: 10.1111/1751-2980.12046. PMID 23419063
- [Background] Chande N, MacDonald JK, McDonald JW. Interventions for treating microscopic colitis: a Cochrane Inflammatory Bowel Disease and Functional Bowel Disorders Review Group systematic review of randomized trials. Am J Gastroenterol. 2009 Jan;104(1):235-41; quiz 234, 242. doi: 10.1038/ajg.2008.16. PMID 19098875
- [Background] Colussi D, Salari B, Stewart KO, Lauwers GY, Richter JR, Chan AT, Ricciardiello L, Khalili H. Clinical characteristics and patterns and predictors of response to therapy in collagenous and lymphocytic colitis. Scand J Gastroenterol. 2015;50(11):1382-8. doi: 10.3109/00365521.2015.1050692. Epub 2015 May 21. PMID 25997458
- [Background] Jarnerot G, Hertervig E, Granno C, Thorhallsson E, Eriksson S, Tysk C, Hansson I, Bjorknas H, Bohr J, Olesen M, Willen R, Kagevi I, Danielsson A. Familial occurrence of microscopic colitis: a report on five families. Scand J Gastroenterol. 2001 Sep;36(9):959-62. doi: 10.1080/003655201750305486. PMID 11521987
- [Background] Kao KT, Pedraza BA, McClune AC, Rios DA, Mao YQ, Zuch RH, Kanter MH, Wirio S, Conteas CN. Microscopic colitis: a large retrospective analysis from a health maintenance organization experience. World J Gastroenterol. 2009 Jul 7;15(25):3122-7. doi: 10.3748/wjg.15.3122. PMID 19575491
- [Background] Khan MA, Brunt EM, Longo WE, Presti ME. Persistent Clostridium difficile colitis: a possible etiology for the development of collagenous colitis. Dig Dis Sci. 2000 May;45(5):998-1001. doi: 10.1023/a:1005593628991. No abstract available. PMID 10795766
- [Background] LaSala PR, Chodosh AB, Vecchio JA, Schned LM, Blaszyk H. Seasonal pattern of onset in lymphocytic colitis. J Clin Gastroenterol. 2005 Nov-Dec;39(10):891-3. doi: 10.1097/01.mcg.0000180634.84689.c2. PMID 16208113
- [Background] Yao MD, von Rosenvinge EC, Groden C, Mannon PJ. Multiple endoscopic biopsies in research subjects: safety results from a National Institutes of Health series. Gastrointest Endosc. 2009 Apr;69(4):906-10. doi: 10.1016/j.gie.2008.05.015. Epub 2009 Jan 10. PMID 19136110